CLINICAL TRIAL: NCT00474305
Title: Effectiveness of Virtual Reality for Persons With PTSD Following a Bus Bombing
Brief Title: Virtual Reality Prolonged Exposure (PE) for Bus Bomb Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: University of Haifa (Other)
Responsible Party: Dr Rena Cooper, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VR-PTSD-HMO-CTIL
Record Dates: First submitted 2007-05-15; First posted 2007-05-16 (Estimated); Last update posted 2010-12-16 (Estimated); Status verified 2010-05

CONDITIONS: PTSD
Keywords: PTSD; Prolonged Exposure; Virtual Reality
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Virtual Reality Treatment for PTSD — 12 session protocol for Prolonged Exposure with Virtual Reality. All sessions 90 minutes.

SUMMARY:
This study will examine whether the use of a Virtual World will be effective in helping treat Posttraumatic Stress Disorder (PTSD). This is a pilot study, with five victims of bus bombings who have developed PTSD. The study will examine pre- and post-treatment levels of PTSD, anxiety, depression and day-to-day functioning.

DETAILED DESCRIPTION:
PTSD can be a long-term debilitating psychiatric problem, occurring following exposure to a traumatic event. Recent studies have shown that Cognitive Behavioral Therapy is effective in the treatment of PTSD. More specifically, a protocol called Prolonged Exposure, where the patient is gradually exposed to feared stimuli, along with building a narrative of the traumatic event, has been shown to reduce PTSD and depression symptoms, both at the end of therapy (9-12 weeks) and at long term follow up.

Despite this success, some patients do not show symptom reduction with this therapy. Virtual Reality, where a real-time virtual world is created, has been successfully used to treat a variety of fears, from pain management to fear of flying. This technique has also been successfully used with patients who have not benefited from Prolonged Exposure for their PTSD, following 9/11.

This study will examine the use of a virtual reality world that involves a bus bombing. It has been created using different levels of exposure to distressing detail, such that the therapist can control the amount of exposure. The protocol is based on Prolonged Exposure, with the Virtual Reality being used to help the patient build a narrative of the event.

Five patients with PTSD following a bus bombing will be treated. They will be assessed pre and post-treatment for symptoms levels of PTSD, depression, anxiety and daily functioning. The treatment consists of 9 sessions, each lasting 90 minutes. Therapy will be supervised, and protocol adherence will be checked by an external therapist. All therapists are trained as supervisors in Prolonged Exposure.

ELIGIBILITY:
Inclusion Criteria:

* PTSD following a bus bombing
* Hebrew speaking

Exclusion Criteria:

* Other psychiatric illness
* Other concurrent intervention

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2007-12; Primary Completion 2011-08 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale (CAPS) | Pre and Post Treatment

SECONDARY OUTCOMES:
Beck Depression Inventory | Pre and Post Treatment
Activity Card Sort | Pre and Post Treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sara A Freedman, PhD, Study Director — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Difede J, Cukor J, Patt I, Giosan C, Hoffman H. The application of virtual reality to the treatment of PTSD following the WTC attack. Ann N Y Acad Sci. 2006 Jul;1071:500-1. doi: 10.1196/annals.1364.052. PMID 16891607
- [Derived] Freedman SA, Hoffman HG, Garcia-Palacios A, Tamar Weiss PL, Avitzour S, Josman N. Prolonged exposure and virtual reality-enhanced imaginal exposure for PTSD following a terrorist bulldozer attack: a case study. Cyberpsychol Behav Soc Netw. 2010 Feb;13(1):95-101. doi: 10.1089/cyber.2009.0271. PMID 20528299